CLINICAL TRIAL: NCT01447290
Title: Comparison of Random Spot Urine Protein:Creatinine Ratio to 24-Hour Timed Urine Protein Collection in the Evaluation of Preeclampsia
Acronym: P:C Ratio
Status: Completed | Type: Observational
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: FWH20110165H
Record Dates: First submitted 2011-10-04; First posted 2011-10-06 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Preeclampsia
Keywords: preeclampsia; protein; creatinine; protein:creatinine ratio
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women being evaluated for preeclampsia

SUMMARY:
This is a non-inferiority, prospective study of the relationship between the 24-hour urine protein collection and spot protein:creatinine ratio in the diagnosis of preeclampsia involving a sample of 18-45 year-old pregnant women attending the new Obstetrics orientation. The investigators will follow all participants who consent to be part of this study throughout their entire pregnancy. Those who get evaluated for preeclampsia will then have a P:C ratio anytime their Primary Obstetrics provider orders a standard of care 24-hour urine collection (standard of care). Those participants who are not evaluated for preeclampsia during their pregnancy will be dropped from the study.

Participants evaluated for preeclampsia during the prenatal period will be asked to provide a random spot clean-catch urine sample at intervals of approximately 0 and 24 hours following the initiation of the 24-hour urine collection. The patient's demographic and clinical data, as well as the spot protein:creatinine ratio and 24-hour urine protein will be collected and analyzed at the conclusion of the study period.

DETAILED DESCRIPTION:
The investigators will recruit a total of 12,000 pregnant female subjects ages 18-45 that have a confirmed positive pregnancy test and whom are attending the new Obstetrics Orientation class. Subjects will be recruited from the MOFH and Eglin.

Visit 1:

* Obtain signed Informed Consent document and HIPAA Authorization (research-driven)
* Review Medical History and record patients age, gestational age, parity and presence of high-risk antepartum conditions (i.e. chronic hypertension, gestational diabetes mellitus-all classes, and pre-existing renal disease) (standard of care)

All participants who consent to be part of this study will be followed throughout their entire pregnancy (birth of child). Those who are identified by their primary obstetrics provider as potentially having preeclampsia will then have a P:C Ratio anytime their Primary Obstetrics provider orders a standard of care 24-hour urine collection (see Antepartum Visit Schedule Below). Those participants who are not evaluated for preeclampsia during their pregnancy will be dropped from the study at the end of their pregnancy (birth of child).

Antepartum Visit:

* Collect 24-hour protein urine (standard of care)
* Collect spot random urine protein:creatinine ratio (at 0 and 24 hours) (research-driven)
* Perform a urinalysis to identify subjects that may have a Urinary Tract Infection (UTI) (if participant tests positive for a UTI, they will be excluded from this data point, however, they will continue in the study and data will be collected from their subsequent urine collections given that the UTI is no longer present) (research-driven)

Participants will be recruited from the new Obstetrics Orientation class so that baseline data may be used to compare a participant's "non-pregnant" physiological state to later gestations (i.e. before and during the time they develop preeclampsia). Previous studies do not directly compare baseline and later gestational data that would show whether the correlation between the P:C ratio and 24 hour urine protein changes or remains unchanged. This data would be more clinically relevant when determining presence of preeclampsia with the understanding that the spot protein:creatinine ratio may or may not retain a strong correlation to the 24 hour urine protein during all gestational ages.

Participants will be continually followed by their Primary Obstetric provider, who will provide standard of care. This includes notifying patients of worsening conditions of preeclampsia, laboratory results, all treatment for preeclampsia, and all teaching involved in the diagnosis and treatment of preeclampsia.

The amount of urine collected for the standard of care 24-hour urine is approximately 2,000 milliliters (mls) of urine. The amount needed in order to process a P:C Ratio is approximately 10mls at 0 hours and 24 hours (total of 20mls).

Participants will follow the standard procedures for a 24-hour urine collection. During the first urination (0 hours) and the last urination (24 hours) participants will pour off 50 mls into a urine cup

Each site's Laboratory will be responsible for analyzing urine samples obtained at their site for this study. Samples will be labeled as they would for standard laboratory draws. All Laboratories are Clinical Laboratory Improvement Amendments (CLIA) certified and will use these procedures when processing Laboratory specimens mentioned in this research project.

SUBJECTS COMPLETING THE STUDY:

Subject's participation in this study is completed at the conclusion of their pregnancy. Subjects will be told the results of their protein urine and spot random urine protein:creatinine ratio by their primary obstetrics provider after each study is completed. Upon completion of the study, each Associate Investigator will send the de-identified data to the Principal Investigator via an encrypted email for analysis. Associate Investigators are also responsible for sending the Principal Investigator all the Informed Consent and HIPAA Authorization documents via encrypted email for retention the conclusion of the study.

WITHDRAWAL PROCEDURES:

If at any time during the study, the subject decides to withdraw from the study, they may do so with no further testing required, beyond that required by standard of care.

DEVIATIONS:

Deviations that do not increase the risks to subjects like those listed in the "risks" section of this protocol are to be reported to the Principal Investigator of this study the 1st workday of every month via the "WHMC Tracking Log for Problems Not Requiring Immediate Reporting". This is done to ensure ongoing monitoring and identification of trends that may arise.

ELIGIBILITY:
Inclusion Criteria:

* Tricare beneficiaries receiving care at Nellis AFB
* Pregnant women (Active Duty Military or DoD beneficiaries) ages 18-45

Exclusion Criteria: None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 18-45 year-old pregnant women (Active Duty Military or DoD beneficiaries) attending the new Obstetrics Orientation class.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with preeclampsia with the protein:creatinine ratio test | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Snyder, D.O., Maj, Principal Investigator — Mike O'Callaghan Military Hospital
Locations (1):
- Michael O'Callaghan Federal Hospital/Nellis Air Force Base, Nellis Air Force Base, Nevada, United States